CLINICAL TRIAL: NCT04931771
Title: Fractional Flow Reserve or 3D-Quantitative-Coronary-Angiography Based Vessel-FFR Guided Revascularization
Acronym: FAST III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ECRI bv (Industry)
Collaborators: Siemens Healthineers AG (Unknown); Pie Medical Imaging (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECRI-15
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Intermediate coronary lesion; Coronary physiology; vFFR
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vFFR guided revascularization (Experimental)
  Interventions: Device: vFFR guided revascularization
- FFR guided revascularization (Active Comparator)
  Interventions: Device: FFR guided revascularization

INTERVENTIONS:
Device: vFFR guided revascularization — 3D-angio-based vessel FFR (CAAS, Pie Medical Imaging, Maastricht, The Netherlands) uses 3-Dimensional Quantitative Coronary Angiography (3D-QCA) for functional assessment of coronary stenosis. vFFR is calculated using two angiographic views with at least 30 degrees difference in rotation/angulation to generate the 3D reconstruction of the coronary artery.
  Arms: vFFR guided revascularization
Device: FFR guided revascularization — Fractional flow reserve (FFR) is a technique used in coronary catheterization to measure pressure differences across a coronary artery stenosis (narrowing, usually due to atherosclerosis) to determine the likelihood that the stenosis impedes oxygen delivery to the heart muscle (myocardial ischemia)
  Arms: FFR guided revascularization

SUMMARY:
The FAST III is a randomized controlled, open-label, multicenter, international, non-inferiority, strategy trial. A total of 2228 participants will be randomized in a 1:1 fashion to either vFFR- or FFR guided revascularization. Patients will be consented prior to the procedure and then followed up to 12 (+1) months after randomization. The primary endpoint is analyzed at 12 months after randomization. Approximately 35 sites in 7 European countries (Netherlands, Ireland, United Kingdom, Germany, Italy, Spain, and France).

DETAILED DESCRIPTION:
The FAST III is a randomized controlled, open-label, multicenter, international, non-inferiority, strategy trial of a vFFR guided strategy as compared to a FFR guided strategy to guide coronary revascularization in 2228 subjects with intermediate coronary artery lesions.

Patients are screened for inclusion/exclusion criteria after the indication for coronary catheterization is established. After providing informed consent, patients are enrolled. Randomization is performed in the randomization module of the EDC system with an allocation ratio of 1:1 and stratification by center. The primary endpoint is a composite of all-cause death, any myocardial infarction, or any revascularization at 1 year post-randomization.

All deaths and major cardiovascular events, including the individual components of primary and secondary endpoints are adjudicated by an independent Clinical Events Committee (CEC), using standardized definitions. An independent Data and Safety Monitoring Board (DSMB) will formally review the accumulating data to ensure there is no avoidable increased risk for harm to participants. The FAST III trial is performed in accordance with the Declaration of Helsinki, Good Clinical Practice (GCP), ISO 14155:2020, EC requirements and country specific regulations.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years of age
2. Presenting with silent ischemia, stable angina, or non-ST-elevation acute coronary syndrome (NSTE-ACS)
3. Coronary artery disease with at least one native artery in which the stenosis severity is questionable (typically 30-80% stenosis)
4. FFR assessment and vFFR assessment feasible
5. The patient is willing and able to cooperate with study procedures and follow-up until study completion
6. Subject is able to confirm understanding of risks, benefits and treatment alternatives and he/she provides informed consent prior to any protocol-related procedure, as approved by the appropriate Ethics Committee

Exclusion Criteria:

1. ST-elevation myocardial infarction (STEMI) at presentation
2. Cardiogenic shock or severe hemodynamic instability at the time of intervention (heart rate<50 beats per minute, systolic blood pressure <90mmHg) or use of left ventricular assist device
3. Any target vessel with a distal Thrombolysis In Myocardial Infarction (TIMI) flow <3.
4. Presence of thrombus in intermediate target lesion.
5. Known untreated severe valvular heart disease
6. Target lesion is located in or supplied by an arterial or venous bypass graft
7. History of cardiac allograft transplantation
8. Aorto-ostial lesions with an estimated diameter stenosis >50%
9. Severe tortuosity precluding the acquisitions of 2 orthogonal projections of the target vessel with minimal overlap or foreshortening.
10. Absolute contraindications or allergy that cannot be pre-medicated, to iodinated contrast or adenosine
11. Non-cardiac co-morbidities with a life expectancy less than 1 year
12. Currently participating in another trial that is not yet at its primary endpoint. The patient is not allowed to participate in another investigational device or drug study until the trial primary endpoint time point is achieved and may only be enrolled once in the study
13. Women of childbearing potential who do not have a negative pregnancy test within 24 hours before the procedure
14. Subject belongs to a vulnerable population (per Investigator's judgment) or subject unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2228 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Rate of the composite of all-cause death, any myocardial infarction, or any revascularization | 1 year
  Procedural myocardial infarction (MI) is adjudicated according to the ARC-2 consensus and spontaneous MI according to the 4th Universal definition of MI.

SECONDARY OUTCOMES:
Rate of patient-oriented composite endpoint (POCE) defined as all-cause death, any stroke, any myocardial infarction, and any revascularization | 1 year
Rate of device-oriented composite endpoint (DOCE) defined as the composite of cardiovascular death, target-vessel MI, clinically indicated repeat revascularization of the target lesion | 1 year
Rate of study-oriented composite endpoint (SOCE) defined as the composite of cardiovascular death, study-vessel or target vessel MI, or study-vessel or target vessel revascularization | 1 year
Rate of target-vessel failure defined as a composite of cardiac death, target vessel myocardial infarction, or clinically indicated target-vessel revascularization | 1 year
Rate of target-lesion failure defined as a composite of cardiac death, target vessel myocardial infarction, or clinically indicated target-lesion revascularization | 1 year
Rate of study-vessel failure defined as a composite of cardiac death, study vessel myocardial infarction, or clinically indicated study-vessel revascularization | 1 year
Rate of definite and probable stent thrombosis | 1 year

OTHER OUTCOMES:
Quality of life (QoL) using the Seattle Angina Questionnaire | 1 month and 1 year
Procedural time | Baseline
Total contrast volume | Baseline
Fluoroscopy time | Baseline
Radiation dose | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joost Daemen, MD, PhD, Principal Investigator — Erasmus Medical Center; Ernest Spitzer, MD, Study Director — European Cardiovascular Research Institute
Locations (43):
- France (7):
  - Clinique St Martin, Caen
  - Institut Cardiovasculaire de Grenoble, Grenoble
  - CHU LILLE - Institut Cœur Poumon, Lille
  - Hôpital de la Croix Rousse, hospices civils de lyon, Lyon
  - Hôpital Privé Jacques Cartier, Massy
  - Clinique les Fontaines, Melun
  - Clinique Saint Hilaire, Rouen
- Germany (6):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charité- Campus Benjamin Franklin, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Marienhaus Klinikum, Neuwied
  - SHG Klinik Völklingen, Völklingen
- Ireland (4):
  - Mater Private Cork, Cork
  - Beaumont Hospital, Dublin
  - Mater Private Dublin, Dublin
  - St James Hospital, Dublin
- Italy (9):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - AOU di Ferrara (Ospedale Sant'Anna), Cona
  - Cardiologia Ospedale Dell' Angelo, Mestre
  - Humanitas Research Hospital, Milan
  - Policlinico San Donato, Milan
  - Pineta Grande Hospital, Naples
  - Ospedale Maggiore della Carità, Novara
  - AOU Verona, Verona
  - Cardiologia Ospedale San Bortolo, Vicenza
- Netherlands (5):
  - Tergooi MC, Blaricum
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer, Dordrecht
  - Erasmus University Medical Center, Rotterdam
  - UMCU, Utrecht
- Spain (8):
  - Hospital Univeritario A Coruna, A Coruña
  - Hospital Clinic, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario de Leon, León
  - Hospital Universitario de la Princesa, Madrid
  - La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clinico Universitario de Valladolid, Valladolid
- United Kingdom (4):
  - Royal Victoria Hospital, Belfast
  - Royal Sussex County Hospital, Brighton
  - Golden Jubilee National Hospital, Glasgow
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scoccia A, Byrne RA, Banning AP, Landmesser U, Van Belle E, Amat-Santos IJ, Sabate M, Tijssen JGP, Spitzer E, Daemen J. Fractional flow reserve or 3D-quantitative-coronary-angiography based vessel-FFR guided revascularization. Rationale and study design of the prospective randomized fast III trial. Am Heart J. 2023 Jun;260:1-8. doi: 10.1016/j.ahj.2023.02.003. Epub 2023 Feb 14. PMID 36796573